CLINICAL TRIAL: NCT05946941
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Deucravacitinib in Adults With Active Sjögren's Syndrome (POETYK SjS-1)
Brief Title: A Study to Evaluate the Efficacy and Safety of Deucravacitinib in Adults With Active Sjögren's Syndrome
Acronym: POETYK SjS-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-1069; 2023-503327-26 (Registry Identifier: EU Clinical Trial Number); U111-1289-6072 (Registry Identifier: WHO)
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Sjögren's Syndrome
Keywords: Deucravacitinib; Sjogren's Syndrome; BMS-986165; POETYK; Sjogren Syndrome; Sjogren-Larson Syndrome; Gougerot-Sjogren; Gougerot Sjogren Syndrome; Sjogren; Sjogren's; Sjogren Disease; Sjogren's Disease
MeSH Terms: conditions — Sjogren's Syndrome | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Deucravacitinib, Dose 1 (Experimental)
  Interventions: Drug: Deucravacitinib
- Deucravacitinib, Dose 2 (Experimental)
  Interventions: Drug: Deucravacitinib
- Placebo, followed by Deucravacitinib Dose 1 or Dose 2 (Placebo Comparator)
  Interventions: Drug: Deucravacitinib; Other: Placebo

INTERVENTIONS:
Drug: Deucravacitinib — Specified dose on specified days
  Other Names: BMS-986165
Other: Placebo — Specified dose on specified days
  Arms: Placebo, followed by Deucravacitinib Dose 1 or Dose 2

SUMMARY:
The purpose of this study is to assess the safety and efficacy of two doses of Deucravacitinib in adult participants with Active Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria

* Satisfy the 2016 American College of Rheumatology/European League Against Rheumatism criteria for the classification of SjS at screening (score ≥ 4), and who have disease duration (from time of initial clinical SjS diagnosis) of at least 16 weeks prior to screening.
* Have moderate to severe SjS ESSDAI ≥ 5.
* Short duration of disease (≤ 10 years) before screening.
* A stimulated whole salivary flow (SWSF) ≥ 0.05 mililiters/minute (mL/minute).
* Positive anti-Sjögren's syndrome-associated antigen A (anti-Ro/SSA) at screening.

Exclusion Criteria

* Autoimmune disease other than SjS (for example, rheumatoid arthritis, systemic lupus erthrematosus [SLE], systemic sclerosis).
* Active fibromyalgia with pain symptoms or signs that would interfere with joint assessment or requiring adjustment in medication within the 3 months before screening to control symptoms; participants with fibromyalgia that is well controlled on stable treatment may otherwise be considered.
* Medical condition associated with sicca syndrome.
* Previous exposure to tyrosine kinase 2 (TYK2) inhibitors such as deucravacitinib or related compounds.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2028-11-16 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) Score at Week 52 | Baseline, Week 52

SECONDARY OUTCOMES:
Change from baseline in European League Against Rheumatism Sjögren's Syndrome Patient Reported Index (ESSPRI) Score at Week 52 | Baseline, Week 52
Number of participants with decrease in ESSPRI ≥ 1 or 15% from baseline at Week 52 | Baseline, Week 52
Number of participants with decrease in ESSDAI ≥ 3 points from baseline at Week 52 | Baseline, Week 52
Number of participants with ESSDAI < 5 at Week 52 | Baseline, Week 52
Change from baseline in ESSDAI at Week 24 | Baseline, Week 24
Change from baseline in stimulated whole salivary flow (SWSF) at Week 52 | Baseline, Week 52
Change from baseline in physician global assessment (PhGA) at Week 52 | Baseline, Week 52
Change from baseline in functional assessment of chronic illness therapy (FACIT)-fatigue at Week 52 | Baseline, Week 52
Change from baseline in ocular dryness numeric rating scale (NRS) at Week 52 | Baseline, Week 52
Change from baseline in oral dryness NRS at Week 52 | Baseline, Week 52
Change from baseline in joint/ muscle pain NRS at Week 52 | Baseline, Week 52
Number of participants with an increase of Schirmer's test ≥ 5 mm if abnormal baseline or no change of Schirmer's test to abnormal if baseline is normal | Baseline, Week 52
Number of participants with adverse events (AEs) | Up to Week 160
Number of participants with serious AEs (SAEs) | Up to Week 160
Number of participants with AEs leading to discontinuation of treatment and study discontinuation | Up to Week 160
Number of participants with AEs of special interest (AESIs) | Up to Week 160
Number of participants with clinical laboratory abnormalities | Up to Week 160
Number of participants with electrocardiogram (ECG) abnormalities | Up to Week 156
Number of participants with vital sign abnormalities | Up to Week 160

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (229):
- United States (31):
  - Local Institution - 0228, Fullerton, California
  - Local Institution - 0222, La Palma, California
  - Local Institution - 0218, San Francisco, California
  - Local Institution - 0203, Santa Monica, California
  - Local Institution - 0067, Denver, Colorado
  - Local Institution - 0049, Clearwater, Florida
  - GNP Research, Cooper City, Florida
  - Local Institution - 0223, Sarasota, Florida
  - Local Institution - 0140, Augusta, Georgia
  - Local Institution - 0229, Lawrenceville, Georgia
  - Local Institution - 0174, Skokie, Illinois
  - Local Institution - 0016, Kansas City, Kansas
  - Local Institution - 0123, Hopkinsville, Kentucky
  - Local Institution - 0017, Baton Rouge, Louisiana
  - Local Institution - 0125, Monroe, Louisiana
  - Local Institution - 0187, Baltimore, Maryland
  - Local Institution - 0173, Boston, Massachusetts
  - Local Institution - 0131, Eagan, Minnesota
  - Local Institution - 0138, Summit, New Jersey
  - Local Institution - 0009, Albuquerque, New Mexico
  - Local Institution - 0184, Mineola, New York
  - Local Institution - 0224, Salisbury, North Carolina
  - Local Institution - 0132, Corvallis, Oregon
  - Local Institution - 0130, Duncansville, Pennsylvania
  - Local Institution - 0022, Jackson, Tennessee
  - Local Institution - 0144, Allen, Texas
  - Local Institution - 0227, Katy, Texas
  - Local Institution - 0175, Plano, Texas
  - Local Institution - 0225, The Woodlands, Texas
  - Local Institution - 0133, Seattle, Washington
  - Local Institution - 0189, Spokane, Washington
- Argentina (10):
  - Local Institution - 0050, San Isidro, Alabama
  - Local Institution - 0100, CABA, Buenos Aires
  - Local Institution - 0003, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0019, Quilmes, Buenos Aires
  - Local Institution - 0026, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0058, Buenos Aires
  - Local Institution - 0137, CABA
  - Local Institution - 0109, City of Buenos Aires
  - Local Institution - 0061, Córdoba
  - Local Institution - 0039, Córdoba
- Australia (2):
  - Local Institution - 0120, Woodville South, South Australia
  - Local Institution - 0165, Nedlands, Western Australia
- Austria (2):
  - Local Institution - 0117, Graz
  - Local Institution - 0087, Vienna
- Belgium (2):
  - Local Institution - 0183, Aalst
  - Local Institution - 0172, Ghent
- Brazil (6):
  - Local Institution - 0170, Vitória, Espírito Santo
  - Local Institution - 0106, Belo Horizonte, Minas Gerais
  - Local Institution - 0091, Juiz de Fora, Minas Gerais
  - Local Institution - 0055, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0018, São Paulo, São Paulo
  - Local Institution - 0111, Uberlândia
- Bulgaria (2):
  - Local Institution - 0008, Plovdiv
  - Local Institution - 0221, Sofia
- Canada (4):
  - Local Institution - 0134, Vancouver, British Columbia
  - Local Institution - 0063, Toronto, Ontario
  - Local Institution - 0004, Sherbrooke, Quebec
  - Local Institution - 0056, Trois-Rivières, Quebec
- Chile (9):
  - Local Institution - 0103, Valdivia, Los Ríos Region
  - Local Institution - 0136, Santiago, Providencia
  - Local Institution - 0032, Viña del Mar, Región de Valparaíso
  - Local Institution - 0097, Santiago, Santiago Metropolitan
  - Local Institution - 0015, Santiago de Chlie, Santiago Metropolitan
  - Local Institution - 0099, Osorno
  - Local Institution - 0121, Santiago
  - Local Institution - 0216, Santiago
  - Local Institution - 0200, Valdivia
- China (32):
  - Local Institution - 0153, Beijing, Beijing Municipality
  - Local Institution - 0156, Beijing, Beijing Municipality
  - Local Institution - 0160, Beijing, Beijing Municipality
  - Local Institution - 0096, Chongqing, Chongqing Municipality
  - Local Institution - 0155, Xiamen, Fujian
  - Local Institution - 0095, Guangzhou, Guangdong
  - Local Institution - 0212, Shenzhen, Guangdong
  - Local Institution - 0180, Luoyang, Henan
  - Local Institution - 0214, Zhengzhou, Henan
  - Local Institution - 0149, Wuhan, Hubei
  - Local Institution - 0094, Changsha, Hunan
  - Local Institution - 0158, Changsha, Hunan
  - Local Institution - 0098, Baotou Shi, Inner Mongolia
  - Local Institution - 0150, Hohhot, Inner Mongolia
  - Local Institution - 0215, Nanjing, Jiangsu
  - Local Institution - 0159, Nanjing, Jiangsu
  - Local Institution - 0154, Suzhou, Jiangsu
  - Local Institution - 0163, Jiujiang, Jiangxi
  - Local Institution - 0177, Nanchang, Jiangxi
  - Local Institution - 0213, Nanchang, Jiangxi
  - Local Institution - 0162, Pingxiang, Jiangxi
  - Local Institution - 0101, Xi'an, Shaanxi
  - Local Institution - 0182, Taiyuan, Shan1xi
  - Local Institution - 0102, Shanghai, Shanghai Municipality
  - Local Institution - 0151, Shanghai, Shanghai Municipality
  - Local Institution - 0157, Shanghai Shi, Shanghai Sheng
  - Local Institution - 0178, Chengdu, Sichuan
  - Local Institution - 0179, Ürümqi, Xinjiang Sheng
  - Local Institution - 0181, Hangzhou, Zhejiang
  - Local Institution - 0152, Hangzhou, Zhejiang
  - Local Institution - 0161, Ningbo, Zhejiang
  - Local Institution - 0093, Wenzhou, Zhejiang
- Colombia (3):
  - Local Institution - 0168, Barranquilla, Atlántico
  - Local Institution - 0043, Chía, Cundinamarca
  - Local Institution - 0037, Bogota D.C
- Denmark (2):
  - Local Institution - 0186, Aarhus, Region Midt
  - Local Institution - 0006, Glostrup Municipality
- Finland (3):
  - Local Institution - 0199, Helsinki
  - Local Institution - 0135, Kuopio
  - Local Institution - 0119, Turku
- France (10):
  - Local Institution - 0072, Orléans, Centre-Val de Loire
  - Local Institution - 0005, Amiens
  - Local Institution - 0073, Bordeaux
  - Local Institution - 0070, Grenoble
  - Local Institution - 0074, Le Havre
  - Local Institution - 0167, Le Kremlin-Bictre
  - Local Institution - 0078, Marseille
  - Local Institution - 0025, Paris
  - Local Institution - 0107, Paris
  - Local Institution - 0057, Paris
- Germany (6):
  - Local Institution - 0079, Munich, Bavaria
  - Local Institution - 0092, Berlin
  - Local Institution - 0031, Freiburg im Breisgau
  - Local Institution - 0033, Hamburg
  - Local Institution - 0075, Tübingen
  - Local Institution - 0051, Würzburg
- Greece (3):
  - Local Institution - 0052, Athens
  - Local Institution - 0077, Athens
  - Local Institution - 0108, Larissa
- Hungary (4):
  - Local Institution - 0115, Budapest, IX, Válassz Egy Opciót…
  - Local Institution - 0113, Budapest
  - Local Institution - 0083, Debrecen
  - Local Institution - 0090, Gyula
- Israel (2):
  - Local Institution - 0145, Ramat Gan, IA
  - Local Institution - 0142, Kfar Saba
- Italy (8):
  - Local Institution - 0065, Brescia
  - Local Institution - 0029, Milan
  - Local Institution - 0124, Napoli
  - Local Institution - 0082, Padua
  - Local Institution - 0128, Pisa
  - Local Institution - 0069, Rome
  - Local Institution - 0062, Rome
  - Local Institution - 0081, Udine
- Japan (26):
  - Local Institution - 0146, Nagoya, Aichi-ken
  - Local Institution - 0205, Toyoake-shi, Aichi-ken
  - Local Institution - 0148, Kitakyushu-shi, Fukuoka
  - Local Institution - 0122, Sapporo, Hokkaido
  - Local Institution - 0188, Sapporo, Hokkaido
  - Local Institution - 0211, Nishinomiya-shi, Hyōgo
  - Local Institution - 0193, Tsukuba, Ibaraki
  - Local Institution - 0202, Kahoku-gun, Ishikawa-ken
  - Local Institution - 0118, Kanazawa, Ishikawa-ken
  - Local Institution - 0206, Kawasaki-shi, Kanagawa
  - Local Institution - 0191, Yokohama, Kanagawa
  - Local Institution - 0139, Sendai, Miyagi
  - Local Institution - 0147, Nagasaki, Nagasaki
  - Local Institution - 0129, Sasebo, Nagasaki
  - Local Institution - 0207, Kurashiki, Okayama-ken
  - Local Institution - 0198, Ōtsu, Shiga
  - Local Institution - 0194, Hamamatsu, Shizuoka
  - Local Institution - 0195, Shimotsugagun, Tochigi
  - Local Institution - 0210, Bunkyo-ku, Tokyo
  - Local Institution - 0196, Bunkyo-ku, Tokyo
  - Local Institution - 0190, Chuo-ku, Tokyo
  - Local Institution - 0201, Meguro-ku, Tokyo
  - Local Institution - 0208, Meguro-ku, Tokyo
  - Local Institution - 0204, Shinagawa-ku, Tokyo
  - Local Institution - 0197, Shinjuku, Tokyo
  - Local Institution - 0192, tabashi City, Tokyo
- Mexico (5):
  - Local Institution - 0020, León, Guanajuato
  - Local Institution - 0023, Guadalajara, Jalisco
  - Local Institution - 0048, Guadalajara, Jalisco
  - Local Institution - 0169, Mexico City, Mexico City
  - Local Institution - 0021, Chihuahua City
- Netherlands (3):
  - Local Institution - 0046, Leeuwarden, Provincie Friesland
  - Local Institution - 0001, Groningen
  - Local Institution - 0105, Rotterdam
- Peru (3):
  - Local Institution - 0047, Jesus Maria, Lima region
  - Local Institution - 0011, Santiago de Surco, Lima region
  - Local Institution - 0171, Lima
- Poland (13):
  - Local Institution - 0084, Krakow, Lesser Poland Voivodeship
  - Local Institution - 0054, Warsaw, Masovian Voivodeship
  - Local Institution - 0141, Warsaw, Woj. Mazowieckie
  - Local Institution - 0010, Warsaw, Woj. Mazowieckie
  - Local Institution - 0024, Bydgoszcz
  - Local Institution - 0085, Bydgoszcz
  - Local Institution - 0040, Lublin
  - Local Institution - 0089, Poznan
  - Local Institution - 0080, Warsaw
  - Local Institution - 0076, Warsaw
  - Local Institution - 0185, Warsaw
  - Local Institution - 0064, Wroclaw
  - Local Institution - 0036, Wroclaw
- Portugal (2):
  - Local Institution - 0028, Lisbon
  - Local Institution - 0014, Lisbon
- Puerto Rico (2):
  - Local Institution - 0143, San Juan
  - Local Institution - 0127, San Juan
- Romania (4):
  - Local Institution - 0220, Cluj-Napoca, Cluj
  - Local Institution - 0041, Brasov
  - Local Institution - 0219, Bucharest
  - Local Institution - 0104, Iași
- South Korea (4):
  - Local Institution - 0110, Seongdong-gu, Seoul
  - Local Institution - 0042, Gwangju
  - Local Institution - 0126, Seoul
  - Local Institution - 0209, Seoul
- Spain (6):
  - Local Institution - 0038, Mérida, Badajoz
  - Local Institution - 0059, Santander, Cantabria
  - Local Institution - 0114, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Local Institution - 0112, A Coruña
  - Local Institution - 0068, Santiago de Compostela
  - Local Institution - 0071, Seville
- Sweden (2):
  - Local Institution - 0166, Gothenburg
  - Local Institution - 0164, Stockholm
- Switzerland (3):
  - Local Institution - 0066, Basel, Baden-Württemberg
  - Local Institution - 0013, Bern
  - Local Institution - 0034, Sankt Gallen
- Taiwan (5):
  - Local Institution - 0116, Kaohsiung City
  - Local Institution - 0012, Taichung
  - Local Institution - 0002, Taichung
  - Local Institution - 0027, Taipei
  - Local Institution - 0045, Taoyuan
- Turkey (Türkiye) (5):
  - Local Institution - 0035, Yenimahalle, Ankara
  - Local Institution - 0088, Ankara
  - Local Institution - 0007, Antalya
  - Local Institution - 0086, Istanbul
  - Local Institution - 0044, Istanbul
- United Kingdom (5):
  - Local Institution - 0176, Southampton, Hampshire
  - Local Institution - 0053, Newcastle upon Tyne, Tyne and Wear
  - Local Institution - 0217, Wolverhampton, West Midlands
  - Local Institution - 0030, Birmingham
  - Local Institution - 0060, Cannock

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05946941.html